CLINICAL TRIAL: NCT02814682
Title: Elaboration of a Multi-dimensional Indicator of Quality in Palliative Care
Acronym: QUALI-PALLI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 10052; PHRQ0904 (Other: The French Ministry of Health)
Record Dates: First submitted 2016-04-01; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2014-11

CONDITIONS: Terminal Illness; End of Life
Keywords: palliative care; quality; indicator; multi-dimensional
MeSH Terms: conditions — Death

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to elaborate a multi-dimensional indicator of the quality in palliative care for patients of end-of-life.

The study will, as secondary objectives:

* elaborate in a standard manner one set of indicators of organization and inner working of a palliative care setting.
* compare according to these indicators, the qualities of 3 types of palliative care: palliative care unit in hospitals, specified identified bed for palliative care patients and non-specified bed.
* explore the relationship between organizational aspects and results in term of burden.

DETAILED DESCRIPTION:
A multicentric study aims on quality of palliative care and will be conducted in three types of 7 palliative care settings: two hospices, two hospital-based palliative care units and three medical units where a mobile palliative care team intervenes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Patient with serious progressive illness and in terminal phase (life expectancy < 3 months): OMS stage is 3 or 4, regardless of etiology.
* Patient informed their diagnosis or not.
* Hospitalized at the moment of inclusion in one of the following care settings: palliative care unit, identified bed or non-identified bed in a care department of short stay.
* No-oppose to participate to the study, by patients, their families or trusted person.

Exclusion Criteria:

* Patient has difficulties in reading, writing or understanding french language, also their family.
* Hospitalization in the palliative care setting < 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population:
  * Patients on palliative care phase,
  * Family members or other people present beside patients,
  * Caregivers (physicians, nurses) who care patients.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Questionnaire for patients | From date of enrollment until the date of first documented leaving from hospital or date of death, whichever came first, up to 2 years
  A questionnaire has been elaborated beforehand by the study will be answered by patients in order to evaluate quality such as reliability, dimensionality and validity against criterion.
Indicator for medical files | At enrollment
  The indicators have been defined by the study, in order to evaluate quality of medical files, such as completeness and discriminatory capacity.
Indicator for caregivers | From date of enrollment until the date of receiving questionnaire returned by caregiver, up to 2 years
  In order to evaluate quality such as reliability and dimensionality, a questionnaire will be answered by caregivers:
  - the Nursing Stress Scale (NSS).
Questionnaire for families | From date of enrollment until the date of receiving questionnaire sent by family, up to 2 years
  A questionnaire has been elaborated, will be answered by patients' families.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GUIRIMAND, MD, Study Chair — Maison Médicale Jeanne Garnier; Philippe Aegerter, MD, PhD, Study Director — Hôpital Ambroise Paré, AP-HP
Locations (1):
- Maison Médicale Jeanne Garnier, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guirimand F, Martel-Samb P, Guy-Coichard C, Picard S, Devalois B, Copel L, Abel A, Ghadi V; QUALI-PALLI group and Philippe Aegerter. Development and validation of a French questionnaire concerning patients' perspectives of the quality of palliative care: the QUALI-PALLI-Patient. BMC Palliat Care. 2019 Feb 11;18(1):19. doi: 10.1186/s12904-019-0403-z. PMID 30744627